CLINICAL TRIAL: NCT06324734
Title: Assessment of Safety of Olaparib in Chinese Patients With Ovarian Cancer in the Real-World Setting
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00082
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Using NCID Database to Assess the Safety of Olaparib in Chinese Patients With Ovarian Cancer by Examining the Incidence, Seriousness, and Severity of All AE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Study D0817R00081 is a retrospective study using NCID database to assess the safety of Olaparib in Chinese patients with ovarian cancer by examining the incidence, seriousness, and severity of all AEs, including but not limiting to AESIs and SAEs, AEs related to Olaparib, and AEs leading to dose reduction, interruption or discontinuation of Olaparib. The first Olaparib prescription date will be set as the index date. The baseline period is from the patient's first ovarian cancer diagnosis recorded in the database to the patient's first treatment with Olaparib (as early as the database start date of January 1, 2013) to the index date for derivation of lines of therapy or one year pre-index date for other baseline variables. Patients will be followed until the patient's last medical record in the database, 30 days after the last dose of Olaparib, death, or June 30, 2023, whichever comes first. All patients who meet the inclusion/exclusion criteria will be enrolled.

DETAILED DESCRIPTION:
Olaparib (Lynparza, formerly referred to as AZD2281 or KU-0059436), is a highly potent polyadenosine diphosphate ribose polymerase (PARP) inhibitor and the first in class approved for use in monotherapy (including maintenance therapy) as well as in combination with other chemotherapeutic agents. It is available in two strengths, 150mg and 100mg. The recommended dosage for Olaparib is 300mg (two 150mg tablets) taken twice daily, resulting in a total daily dose of 600mg. The 100mg strength tablet is used for dose reduction purposes. In August 2018, based on the findings of the trials, Assessment of Efficacy of AZD2281 in Platinum Sensitive Relapsed Serous Ovarian Cancer (Study 19, NCT00753545) and Olaparib Treatment in Breast Cancer Gene (BRCA) Mutated Ovarian Cancer Patients After Complete or Partial Response to Platinum Chemotherapy (SOLO-2, NCT01874353), China National Medical Products Administration (NMPA) approved Olaparib tablets for the maintenance treatment of adult patients with platinum-sensitive recurrent epithelial ovarian cancer, fallopian tube cancer,or primary peritoneal cancer who have achieved a complete or partial response to platinum-bSAEd chemotherapy. In November 2019, based on the results of the trial, Olaparib Maintenance Monotherapy in Patients With BRCA Mutated Ovarian Cancer Following First Line Platinum Based Chemotherapy (SOLO-1, NCT01844986), Olaparib received approval for the maintenance treatment of treatment-naïve adult patients with advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer who have germline BRCA mutations (gBRCAm) or somatic BRCA mutations (sBRCAm) and have achieved a complete or partial response to first-line platinum-based chemotherapy in China. Furthermore, in September 2022, based on the in PAOLA-1 study in front-line advanced ovarian cancer (NCT02477644), Olaparib in combination with Bevacizumab was approved for the maintenance treatment of adult patients with homologous recombination deficiency (HRD)-positive advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer who have achieved a complete or partial response to first-line platinum-based chemotherapy in China. Lynparza has been reported to be associated with mild or moderate adverse reactions [grade 1 or 2 according to the Common Terminology Criteria for Adverse Events (CTCAE)] and generally not requiring treatment discontinuation. In accordance with the Measures for the Administration of Adverse Drug Reaction Reporting and Monitoring (Order No.81 of the Ministry of Health), it is recommended to monitor the safety profile of newly approved drugs in real-world settings. Post-marketing real-world studies closely reflect clinical practice and provide a comprehensive understanding of the product's safety profile compared to premarketing Phase II/III studies. Currently, there is a limited number of safety studies focusing on Chinese patients with ovarian cancer conducted in routine clinical practice, and these studies have small sample size. This study aims to assess the safety of Olaparib in Chinese ovarian cancer patients treated in real-world clinical practice by retrospectively analysing electronic medical records (EMR) of ovarian cancer patients who received Olaparib in China from August 2018 to June 2023, documented in the National Cancer Information Database (NCID).

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed with advanced or platinum sensitive recurrence epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (FIGO stage III-IV) treated with Olaparib+/-Bevacizumab according to approved label indications in China;
2. Patients with at least one prescription record of Olaparib between August 01, 2018 and June 30, 2023;
3. Age ≥18 years at first use of Olaparib;
4. At least one visit record after the first use of Olaparib.

Exclusion Criteria:

* Patients enrolled in the other Olaparib DIM Programs (D0816C00016 and D0817R00011) conducted by AstraZeneca.
* Patients newly diagnosed with stage I and stage II ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (age>=18 years) who were newly diagnosed advanced or platinum sensitive recurrence epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, and used Olaparib（monotherapy or in combination with Bevacizumab in 1L maintenance setting， or monotherapy in PSR setting） during the study timeframe will be included in the study.
  Patients will be excluded if they don't have any visit record post use of Olaparib or they were enrolled in the other Olaparib Intensive Monitoring Studies (D0816C00016 and D0817R00011) conducted by AstraZeneca.
Sampling Method: Non-Probability Sample
Enrollment: 2506 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
The incidence, seriousness, and severity of all AEs | August 1, 2018 to June 30, 2023.
  To assess the safety of Olaparib in Chinese ovarian cancer patients in real-world clinical practice by examining the incidence, seriousness, and severity of all adverse events (AEs), including but not limiting to adverse events of special interest (AESIs), serious adverse events (SAEs), AEs causally related to Olaparib, and AEs leading to dose reduction, interruption, or discontinuation of Olaparib.(classified by 1st Line(1L) 1L Olaparib mono,1L Olaparib
  +Bevacizumab, Platinum Sensitive Recurrence(PSR) Olaparib mono)

SECONDARY OUTCOMES:
The number and proportion of patients according to different baseline demographics and characteristics | August 1, 2018 to June 30, 2023.
  To describe the baseline demographics and clinical characteristics of Chinese ovarian cancer patients treated with Olaparib in real-world clinical practice and to assess the safety of Olaparib in different subgroups. The subgroup analysis will be conducted according to age, comorbidities , gene status，stage, number of lines of chemotherapy, duration of Olaparib treatment, etc.
Overall number and proportion of patients with olaprib combination maintenance therapy in PSR patients | August 1, 2018 to June 30, 2023.
  To describe the baseline demographics and clinical characteristics of Chinese ovarian cancer patients treated with Olaparib in real-world clinical practice and to assess the safety of Olaparib in different subgroups. The subgroup analysis will be conducted according to age, comorbidities , gene status，stage, number of lines of chemotherapy, duration of Olaparib treatment, etc.

OTHER OUTCOMES:
Overall number and proportion of patients with olap arib combination maintenance therapy in 1L patients 2) | August 1, 2018 to June 30, 2023.
  To describe the treatment patterns of Olaparib in Chinese ovarian cancer patients in real-world clinical practice.
  1. proportion of Olaparib combo maintenance therapy(Olaparib+Oral anti-angiogenic therapy
     / Immunotherapy /Other) in1Lpatients
  2. proportion of Olaparib combo maintenance therapy(Olaparib+anti-angiogenic therapy / Immunotherapy /Other)) in PSR patients

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- See also: D0817R00082_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0817R00082&attachmentIdentifier=2bf5b5ec-061d-40a6-b36c-e6c15b2d1aa5&fileName=D0817R00082_CSR_Synopsis_Redacted.pdf&versionIdentifier=